CLINICAL TRIAL: NCT05298293
Title: Evaluation of a Web Application on Event Reporting for Patients With B Lymphoma on First Line Treatment
Brief Title: Electronic MonitorIng of Events for dIffuse Large b Cell LYmphoma
Acronym: EMILY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weprom (Other)
Collaborators: Resilience (Industry); Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: WP-2022-01; 2021-A02957-34 (Other: French Health Products Safety Agency)
Record Dates: First submitted 2022-03-07; First posted 2022-03-28 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: ONCOLAXY web-application; electronic Patient Reported Outcomes
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ONCOLAXY follow-up (Experimental): patients will make a regular assessment of symptoms via an electronic questionnaire
  Interventions: Device: ONCOLAXY Follow-up
- Standard follow-up (No Intervention): patients will have the standard follow-up

INTERVENTIONS:
Device: ONCOLAXY Follow-up — The operation of Oncolaxy© is based on the principle of e-PRO (electronic patient reported outcome) which is able to assess the symptoms declared by patients treated for cancer, to detect an evolution, a recurrence or the toxicity of a therapy. Alerts are sent to the healthcare team if the algorithm detects suspicious symptoms or worsening of these symptoms.
  Oncolaxy© records symptoms using an electronic questionnaire that allows them to be graded. Questionnaires are sent out on a regular basis. The algorithm analyzes the responses and processes them taking into account the score of the response and its evolution over time. The combination of the results makes it possible to send information to the healthcare teams in charge of the patient that will alert them, enlighten them and help them guide their decisions which remain under their sole control. The summary of the results can be viewed at any time on a dashboard.
  Arms: ONCOLAXY follow-up

SUMMARY:
Diffuse large B cell lymphoma is the most common malignant lymphoid hemopathy. More than half of the patients will be cured with an RCHOP-type immunochemotherapy protocol (Rituximab, Cyclophosphamide, Doxorubicin, Vincristine, Prednisone). Monitoring of adverse effects, risk of relapse and quality of life are essential in overall management. Patients are the best candidates to report them. Managing these events should improve quality of life and reduce costs. The aim of this study is to assess the feasibility of monitoring these events by a web application (Oncolaxy©) and to compare it with a control population in the context of a randomized pilot study including 80 patients per arm with diffuse large cell B lymphoma in first-line treatment with R-CHOP.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with untreated large B cell lymphoma requiring a first line treatment by RCHOP or R-mini-CHOP
2. Patient aged 18 years or older at the time of signing Informed Consent Form
3. Additional Intrathecal or/and intravenous treatment with Methotrexate allowed, if indicated
4. Eastern Cooperative Oncology Group (ECOG) Performance Status < 3
5. Patient with internet access (or has someone at home who can help send patients' symptoms or complete the form)
6. Patient enrolled in social security
7. Patient has given his written consent ahead of any specific protocol procedure

Exclusion Criteria:

1. Patient with symptomatic brain metastases,
2. Patient deprived of their liberty, under guardianship or trusteeship
3. Patient is being treated for another cancer and has not been cured
4. Patient with dementia, mental disorders or psychological pathology which could compromise patient informed consent and/or the observance of the study protocol
5. Patient cannot submit to the protocol for psychological, social, familial or geographical reasons
6. Patient is pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Description of events | 29 months
  The events will be collected (CTCAE V5.0) per patient
Delay of taking care of event | 29 months
  The period of management of event will be evaluated between the date of the event and the first action realize to manage this event (patient contact, consultation, hospitalization, prescription, etc.) incremented in the source file
Description of emergency entry | 29 months
  The number of emergency visits (consultation or hospitalization in the suites) per arm
Description of hospitalisations | 29 months
  The number and average length of stay of hospitalizations per patient and per arm
Description of dose/intensity of RCHOP regimen | 29 months
  The dose of treatment received compared to the theoretical dose will assess the dose / intensity
Description of treatment interruptions | 29 months
  The number of patients having had a treatment interruption will be recorded out of the total number of patients
Description of the quality of life | 29 months
  Quality of life will be evaluated by the Quality of Life Questionnaire-C30 (QLQ-C30). QLQ-C30 is a generic questionnaire for cancer patients. Score will be calculated according to EORTC guidelines. The scores range from 0 to 100; a higher score represents a higher ("better") level of functioning, or a higher ("worse") level of symptoms. QoL with QLQ-C30 will be evaluated before start of treatment, at the 3rd cycle, 6th and 8th cycles of treatment and then at 12 and 24 months. Score will be calculated according to EORTC guidelines
Description of anxiety | 29 months
  Anxiety will be evaluated by the State-Trait Anxiety Inventory Form Y (STAI-Y scale). STAI-Y is a specific questionnaire for which reflects the current emotional state (STAI-form Y-A) which makes it possible to assess the nervousness and anxiety of the patient. The scores range from 20 to 80; Higher score is worse.
  STAI-Y will be evaluated before start of treatment, at the 3rd cycle, 6th and 8th cycles of treatment and then at 12 and 24 months.
Description of patient's satisfaction with specific questionnaire dedicated to the use of the web-application | 29 months
  Patient satisfaction will be evaluated by a specific self-evaluation (specific questionnaire dedicated to the use of the web-application) at the end of treatment, 12th and 24th months follow-up visits. The scores range from 14 to 70; Higher score is better.
Overall survival | 29 months
  Overall survival will be calculated from the date of randomization to the date of death due to any cause or the date last known to be alive if patient is censored
Progression Free survival | 29 months
  Progression Free survival will be calculated from the date of randomization to the date of first progression of disease based on Investigator assessment per Lugano classification or the date of death or censored at the date of the last valid tumor assessment
Event-free survival | 29 months
  Event-free survival will be defined as the time between the date of treatment initiation and the date of the first event (relapse, death, unplanned hospitalizations) demonstrated or the date of death if the patient died or the date of the last news if the patient is censored,
Description of health care team satisfaction by a specific questionnaire dedicated to the use of the web-application | 29 months
  Health care team satisfaction will be evaluated by a specific questionnaire (specific questionnaire dedicated to the use of the web-application) at the 6th and 12th of use of application. The scores range from 8 to 33; Higher score is worse.
Description of face-to-face consultations | 29 months
  In the application arm the number of face-to-face consultations triggered by an alert
Description of teleconsultations | 29 months
  In the application arm the number of teleconsultations triggered by an alert
Description of drug prescriptions | 29 months
  In the application arm the number of drug prescription triggered by an alert
Description of nursing prescription | 29 months
  In the application arm the number of nursing prescription triggered by an alert

CONTACTS AND LOCATIONS:
Overall Officials: Katell LE DÛ, MD, Principal Investigator — Hôpital Privée du Confluent
Locations (5):
- France (5):
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - Clinique Victor Hugo/Centre Jean Bernard/ILC, Le Mans
  - Hôpital Privée du Confluent, Nantes
  - Centre Hospitalier de St Nazaire, Saint-Nazaire
  - Centre de radiothérapie de Robertsau, Strasbourg

IPD SHARING:
Plan to Share IPD: No